CLINICAL TRIAL: NCT04849351
Title: A Multi-center, Single-arm, Open-label Clinical Study to Evaluate the Efficacy and Safety of HMPL-689 in Patients With Relapsed/Refractory Marginal Zone Lymphoma and Follicular Lymphoma
Brief Title: Clinical Study of HMPL-689 for Relapsed/Refractory Marginal Zone Lymphoma and Follicular Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-689-00CH3
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Marginal Zone Lymphoma; Follicular Lymphoma
Keywords: Marginal Zone Lymphoma; Follicular Lymphoma; Phosphatidylinositol 3-kinase inhibitor
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Relapsed/Refractory MZL and FL (Experimental): Relapsed/Refractory Marginal Zone Lymphoma and Follicular Lymphoma
  Interventions: Drug: HMPL-689

INTERVENTIONS:
Drug: HMPL-689 — All patients are to receive monotherapy of HMPL-689 30 mg QD continuously in 28-day treatment cycles.
  Other Names: Phosphatidylinositol 3-kinase-δ inhibitor

SUMMARY:
A Multi-center, Single-arm, Open-label Clinical Study to Evaluate the Efficacy and Safety of HMPL-689 in Patients with Relapsed/Refractory Marginal Zone Lymphoma (MZL) and Follicular Lymphoma (FL)

DETAILED DESCRIPTION:
This is a multi-center, single-arm, open-label clinical study to evaluate the oral therapy with HMPL-689 in patients with relapsed / refractory MZL and FL. Relapse / refractory is defined as such a situation when a patient has not achieved response (CR or PR) after the latest line of systemic treatment, or has disease progress (PD) or relapse after achieving response. Two (2) cohorts of patients will be enrolled in this study:

Cohort 1: approximately 81 patients with histologically confirmed MZL

Cohort 2: approximately 104 patients with histologically confirmed FL (pathological grade 1-3a)

All patients are to receive monotherapy of HMPL-689 30 mg once a day (QD) continuously in 28-day treatment cycles until PD / recurrence, patient death, intolerable toxicity, initiation of other antitumor therapy, the patient unable to further benefit from the study treatment as judged by the investigators, the patient or his/her legal representative's request to withdraw from the clinical study treatment, the patient lost to follow-up or end of the study, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Patients with relapsed/refractory marginal zone lymphoma or follicular lymphoma
3. Eastern Cooperative Oncology Group (ECOG) Performance Status score 0-2;
4. At least one measurable lesion by computerised tomography (CT) / magnetic resonance imaging (MRI) (the longest diameter of nodal lesion > 1.5 cm or extranodal lesion > 1 cm);
5. Expected survival of more than 12 weeks;

Exclusion Criteria:

1. Having lymphoma with central nervous system (CNS) or cerebral pia mater invasion;
2. Known histologic transformation to aggressive lymphomas such as diffuse large B-cell lymphoma (DLBCL);
3. Prior use of any phosphatidylinositol 3-kinase (PI3K) inhibitor;
4. Inadequate organ function of liver and kidney;
5. Currently known active infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV);
6. Having received systemic antitumor therapy or radiotherapy within 4 weeks prior to the first dose of the investigational product;
7. Toxicity of previous antitumor therapy not recovered to CTCAE grade ≤ 1, except alopecia, prior to the first dose of the investigational product;
8. Complicated with uncontrolled systemic infection requiring intravenous antibiotic treatment;
9. Pregnant (positive serum pregnancy test) or lactating women;
10. Any other disease, metabolic abnormality, physical examination abnormality or clinically significant laboratory test abnormality, one disease or state providing a reason to suspect that the subject is not suitable for HMPL-689 at the investigator's discretion, or one condition that will affect interpretation of the study results or bring the subject at high risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Baseline up to the last patient has completed 12 months after treatment.
  Defined as the proportion of patients with CR or PR

SECONDARY OUTCOMES:
Complete response (CR) rate | Baseline up to the last patient has completed 12 months after treatment.
  Defined as the proportion of patients with CR.
Progression-free survival (PFS) | Baseline up to the last patient has completed 12 months after treatment.
  Defined as the time from the first dose of HMPL-689 to occurrence of PD or death, whichever comes first.
Time to response (TTR) | Baseline up to the last patient has completed 12 months after treatment.
  Defined as the time from the first dose of HMPL-689 to the first objective response.
Duration of response (DoR) | Baseline up to the last patient has completed 12 months after treatment.
  Defined as the time from the initial objective response to disease recurrence, progression or death.
Overall survival (OS) | Baseline up to the last patient has completed 12 months after treatment.
  Defined as the time from the first dose with HMPL-689 to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: junning Cao, Ph.D, Principal Investigator — Fudan University; Zhiming Li, post-doc, Principal Investigator — Sun Yat-sen University
Locations (58):
- China (58):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Chao-yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing GoBroad Boren Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - Hainan General Hospital, Haikou, Hainan
  - Affiliated Hospital of Chengde Medical University, Chengde, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Hospital of Harbin, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Puyang Oilfield General Hospital, Puyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - People's Hospital of Wuhan University, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second People's Hospital of Huaihua, Huaihua, Hunan
  - The Central Hospital of YongZhou, Yongzhou, Hunan
  - The First People's Hospital of Nantong, Nantong, Jiangsu
  - The Second Affiliated Hospital of Suzhou University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Gannan Medical University, Gannan, Jiangxi
  - Ganzhou People's Hospital, Ganzhou, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jiangxi Provincial Cancer Hospital, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - Shengjing Hospital of China Medical University, Shengyang, Liaoning
  - Affiliated Hospital of Binzhou Medical University, Binzhou, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The affiliated hospital of Qingdao University, Qingdao, Shandong
  - Xinhua Hospital affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Tongji University School of Medicine, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Cancer Hospital Affiliated to Xinjiang Medical University, Ürümqi, Xinjiang
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang